CLINICAL TRIAL: NCT04184700
Title: Epigenetic Effects Involved in Children With Cow's Milk Allergy: A Possible Effect of Hypoallergenic Formulas
Brief Title: Epigenetic Effects in Children With Cow's Milk Allergy Treated With Different Formulas
Acronym: EPICMA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Full professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28n15
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EHCF + LGG (Experimental): Extensively hydrolyzed casein formula plus Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: EHCF+LGG
- RHF (Active Comparator): Extensively hydrolyzed rice formula
  Interventions: Dietary Supplement: RHF
- EHWF (Active Comparator): Extensively hydrolyzed protein formula
  Interventions: Dietary Supplement: EHWF
- AAF (Active Comparator): Amino acid based formula
  Interventions: Dietary Supplement: AAF
- SF (Active Comparator): Soy formula
  Interventions: Dietary Supplement: SF

INTERVENTIONS:
Dietary Supplement: EHCF+LGG — Extensively hydrolyzed casein formula containing Lactobacillus rhamnosus GG
  Arms: EHCF + LGG
Dietary Supplement: RHF — Rice hydrolysed formula
  Arms: RHF
Dietary Supplement: SF — Soy formula
  Arms: SF
Dietary Supplement: EHWF — extensively hydrolysed whey formula
  Arms: EHWF
Dietary Supplement: AAF — amino acid based formula
  Arms: AAF

SUMMARY:
Lactobacillus GG (LGG) is able to exert long lasting effects in children with atopic disorders. Nutramigen LGG accelerates tolerance acquisition in infants with cow's milk allergy. The mechanisms of these effects are still largely undefined. The effect of LGG could be related at least in part by the immunoregulatory role played by LGG. This probiotic can balance the generation of cytokines possibly involved in IgE- or non-IgE-mediated cow's milk allergy Interleulkin (IL)-4, IL-5, IL-10, IFN-γ , TGF-β, and TNF-Υ), which can contribute to modulation of inflammatory processes. The investigators have demonstrated that children with IgE-mediated CMA produce significantly higher level of IL-4 and IL-13 in response to cow's milk protein, and that tolerance is associated with a marked reduction of IL-13 production and a concomitant increased frequency of IFN-γ releasing cells. Epigenetics studies the heritable (and potentially reversible) changes of the genome inherited from one cell generation to the next which alter gene expression but do not involve changes in primary DNA sequences, highlighting the complexity of the inter-relationship between genetics and nutrition. There are three distinct, but closely interacting, epigenetic mechanisms (histone acetylation, DNA methylation, and non-coding microRNAs) that are responsible for modifying the expression of critical genes associated with physiologic and pathologic processes. The profile of epigenetic modifications associated with Th lineage commitment, coupled with the sensitivity of the early developmental period, has led to speculation that factors that disrupt these pathways may increase the risk of allergic diseases. Specifically, effects on DNA methylation and endogenous histone deacetylase inhibitors acting on specific pathways (Th1 and T regulatory cell differentiation) may favour Th2-associated allergic differentiation. MicroRNAs are another structural components of an epigenetic mechanism of post-transcriptional regulation of messenger RNA translation. It has been recently identified a specific Th2-associated microRNA (miR-21) that is critical for the regulation of Th cell polarization. It has been previously demonstrated an inverse DNA methylation pattern of cytokines involved in Th2 response (IL-4, IL-5) compared with cytokines involved in Th1 response (IL-10, INF- y) in children with CMA acquiring oral tolerance, with the most pronounced effects in those treated with Nutramigen LGG.

ELIGIBILITY:
Inclusion Criteria:

* children with cow's milk allergy

Exclusion Criteria:

* Concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protein-induced enterocolitis syndrome,
* suspected cow's milk protein-induced anaphylaxis,
* still on exclusion diet with one of the study formulas or with another dietary regimen because of cow's milk allergy,
* other food allergies.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Epigenetic modifications in cytokines genes | 12 months
  Expression (fc, fold change, ΔΔCt method)) of FOXP3 in children with cow's milk allergy
Epigenetic modifications in cytokines genes | 12 months
  TSDR demethylation rate (%) of FOXP3 in children with cow's milk allergy

SECONDARY OUTCOMES:
microRNAs modifications | 12 months
  Expression of miR-125b miR-146a miR-155 miR-29a/b miR-27a miR-128 miR-21 miR-126 miR-145 miR-106a miR-193a5p miR-128
Concentration of metagenomic characteristics of the intestinal microbiota | 12 months
  evaluation of composition of gut microbiota
Concentration of metabolomic characteristics of the intestinal microbiota | 12 months
  evaluation of function of gut microbiota
The rate of patients with immune tolerance acquisition to cow's milk protein | 12 months
  Rate of patients with acquisition of tolerance to cow milk protein (rate of patients with outgrown cow's milk allergy)
Epigenetic modifications in cytokines genes | 6 and 12 months
  Methylation rate (%) of interleukin IL-4, IL-5, IL-10, IFN-γ, in children with cow's milk allergy
Epigenetic modifications in cytokines genes | 6 and 12 months
  Serum levels (pg/ml) of interleukin IL-4, IL-5, IL-10, IFN-γ in children with cow's milk allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Office, Naples, Italy

IPD SHARING:
Plan to Share IPD: No